CLINICAL TRIAL: NCT02538705
Title: Safety and Efficacy Study of Pl-vegf165 to Treat Diabetic Foot Syndrome
Brief Title: Safety and Efficacy Study of Neovasculgen (Pl-VEGF165) Gene Therapy in Patients With Diabetic Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artgen Biotech (Other)
Collaborators: Ryazan State Medical University (Other); Vidnoe District Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoFoot Pilot Study
Record Dates: First submitted 2015-08-30; First posted 2015-09-02 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2015-08

CONDITIONS: Ulcers Related to Diabetic Foot Syndrome
Keywords: Diabetic foot syndrome; Ulcers
MeSH Terms: conditions — Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neovasculgen (Experimental)
  Interventions: Drug: Neovasculgen

INTERVENTIONS:
Drug: Neovasculgen
  Other Names: pl-vegf165

SUMMARY:
The purpose of this study is to determine whether pl-vegf165 (Neovasculgen) is effective in the treatment of ulcers related to diabetic foot syndrome

DETAILED DESCRIPTION:
This is a open clinical trial assessing the therapeutic efficacy of pl-vegf165 (Neovasculgen) in treating ulcers related to diabetic foot syndrome. Each patient will undergo several intramuscular injections with a treatment dose of pl-vegf165 (Neovasculgen) in calf of affected extrimity.

Study participants at the first study visit will complete study questionnaires, their foots will be assessed clinically for ulceration. After this initial assessment, the patients will undergo intramuscular injections of pl-vegf165 (Neovasculgen) in a calf altered with ulcers due to diabetic foot syndrome.

At three month post-injection, the patient will complete study questionnaires, their foots will be assessed clinically for ulceration, and their foots will undergo non-invasive transcutaneous oximetry measurement. At six months post-injection, the patient will again complete study questionnaires, their foots will be assessed clinically for ulceration and will undergo non-invasive transcutaneous oximetry measurement.

ELIGIBILITY:
Inclusion Criteria:

* obtained voluntary informed consent for participation in the clinical study
* presence of diabetic foot syndrome
* presence at least one active ulcer at baseline

Exclusion Criteria:

* Any disease that can, in the opinion of the treating physician, affect the outcome of the study
* Patients with addictive disorders or substance abuse
* Pregnancy or nursing
* All other exclusion criteria listed in the summary of product characteristics (SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Area of diabetic foot ulcers | 180 days
  To determine the ability of pl-vegf165 to facilitate and accelerate diabetic foot ulcers healing

SECONDARY OUTCOMES:
Transcutaneous oxygen pressure | 180 days
  To determine the ability of pl-vegf165 to improve blood circulation in affected extremity by angiogenesis inducing

CONTACTS AND LOCATIONS:
Locations (1):
- Human Stem Cell Institute, Moscow, Russia